CLINICAL TRIAL: NCT06544161
Title: Measurement of Occlusion Pressure of the External Jugular Vein for Intravascular Volume Assessment in Cirrhotic Patients During Intravenous Albumin Substitution.
Brief Title: EJV Occlusion Pressure Measurement to Assess Intravascular Volume in Cirrhotic Patients During IV Albumin Substitution
Acronym: CPMX2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Compremium AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-D0007
Record Dates: First submitted 2024-07-22; First posted 2024-08-09 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Liver Cirrhosis
Keywords: Cirrhosis; Albumin; Volume overload
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPMX2 Arm (Other): This study is a single-center, single arm, prospective, exploratory proof of concept study.
  Cirrhotic patients with an indication for intravenous albumin will undergo a venous compression technique of the external jugular vein plus an ultrasound examination before/after passive leg raise as well as before/after intravenous albumin infusion in order to study the dynamics of the intravascular volume status and to rule out volume overload.
  Interventions: Device: CPMX2

INTERVENTIONS:
Device: CPMX2 — The CPMX2 is a point-of-care device for non-invasive, real-time, and intermittent monitoring of vascular occlusion pressure.

SUMMARY:
Cirrhotic patients with an indication for intravenous albumin will undergo a venous compression technique of the external jugular vein plus an ultrasound examination before/after passive leg raise as well as before/after intravenous albumin infusion in order to study the dynamics of the intravascular volume status and to rule out volume overload.

DETAILED DESCRIPTION:
Cirrhotic patients with portal hypertension are prone to develop ascites. Current guidelines recommend volume expansion using intravenous (IV) albumin infusion for several circumstances, such as large volume paracentesis, development of spontaneous bacterial peritonitis (SBP), and treatment of acute kidney injury (AKI) with/without hepatorenal syndrome (HRS). However, current dosages for IV albumin infusion do not consider individual intravascular volume status before its administration. In addition, there are increasing reports of volume overload following volume expansion with albumin in cirrhotic patients within and beyond current indications. Non-invasive point-of-care ultrasound (POCUS) of the inferior vena cava (IVC) diameter and collapsibility index (IVCCI) using echocardiography has been proposed for assessing volume status in patients with cardiac disease and for predicting fluid responsiveness in critically ill patients. In addition, determining the occlusion pressure of the external jugular vein (EJV) has been proposed as a surrogate parameter for the estimation of central venous pressure (CVP). In 2005, Baumann et al. introduced a novel method for non-invasive venous pressure measurement by combining ultrasound and a tissue pressure manometer. Peripheral occlusion pressure was measured non-invasively via jugular and basilic vein. Although good correlation with invasive CVP measurements was achieved and measurements showed potential to reflect patients' 'tolerable reserve' with respect to fluid-overload in intensive care and cardiologic patients, its application in cirrhotic patients needs to be studied.

In this study, the investigators aim to assess whether compression of the EJV is feasible in the cirrhotic patients population and observe the change in EJV occlusion pressure determined by the CPMX2 in parallel to sonographic assessment of the IVC diameters and IVCCI as indicators for changes in intravascular volume status in patients with decompensated cirrhosis and an indication for intravenous albumin substitution.

The objective of this clinical investigation is to assess safety and feasibility of external jugular vein (EJV) occlusion pressure measured non-invasively with CPMX2 in patients with decompensated cirrhosis with an indication for albumin infusion.

Data gathered in this study will help define hypotheses to be used in future clinical investigations about the role of absolute values and/or changes in EJV occlusion pressure in characterizing intravascular volume status and its change after passive leg elevation (as an indirect test for fluid responsiveness) and intravenous albumin infusion (for volume expansion) in patients with decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* In- and outpatients with liver cirrhosis of any etiology, diagnosed by either liver histology or compatible biochemical, imaging and clinical parameters, being treated at the department of Visceral Surgery and Medicine at Inselspital Bern, University Hospital Bern, Switzerland.
* Age ≥ 18 years
* Indication for IV albumin infusion according to current EASL guidelines[11] and BAVENO VII consensus recommendations[12] including large volume paracentesis, spontaneous bacterial peritonitis (SBP), AKI with/without HRS.
* Available transthoracic echocardiography assessing right heart function within maximum 3 months from study inclusion.

Exclusion Criteria:

* Patients admitted to intermediate care unit or intensive care unit at the time of albumin infusion
* Previous IV albumin infusion within the last 5 days
* Contraindication to the PLR test (i.e. increased intracranial pressure)
* Contraindication to albumin infusion (i.e. anaphylactic reactions against albumin)
* History of right heart failure
* Clinical evidence of lung edema, hemodynamic instability/shock
* Anatomic IVC abnormalities, such as IVC stenosis and/or thrombosis
* History of orthotopic liver transplant
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Absolute values and relative changes in external jugular vein (EJV) occlusion pressure | Immediately before (10 seconds) and 1 minute after sustained passive leg raising (PLR) as well as immediately before (10 seconds) and after IV albumin infusion (total duration of procedure approximately 2 hours/patient)
  Reporting of absolute values (minimum and maximum mmHG) and relative changes in % in external jugular vein (EJV) occlusion pressure as measured with CPMX2.
Feasibility of using CPMX2 in clinical conditions | During the procedure which should last about 2 hours/patient
  Feasibility of using CPMX2 in clinical conditions will be evaluated through a usability and workflow questionnaire for the practitioner (description).

SECONDARY OUTCOMES:
Absolute values and relative changes in inferior vena cava (IVC) maximal diameter | Immediately before (10 seconds) and 1 minute after sustained passive leg raising (PLR) as well as immediately before (10 seconds) and after IV albumin infusion (total duration of procedure approximately 2 hours/patient)
  Reporting of absolute values and relative changes of the the inferior vena cava (IVC) maximal diameter (in mm) done with point-of-care ultrasound during the specified time frame (description).
Absolute values and relative changes in inferior vena cava (IVC) minimal diameter | Immediately before (10 seconds) and 1 minute after sustained passive leg raising (PLR) as well as immediately before (10 seconds) and after IV albumin infusion (total duration of procedure approximately 2 hours/patient)
  Reporting of absolute values and relative changes of the the inferior vena cava (IVC) minimal diameter (in mm) done with point-of-care ultrasound during the specified time frame (description).
Absolute values and relative changes in inferior vena cava (IVC)-collapsibility index | Immediately before (10 seconds) and 1 minute after sustained passive leg raising (PLR) as well as immediately before (10 seconds) and after IV albumin infusion (total duration of procedure approximately 2 hours/patient)
  Reporting of absolute values and relative changes of the the inferior vena cava (IVC)-collapsibility index (in %) done with point-of-care ultrasound during the specified time frame (description).
Evaluation of preliminary performance of CPMX2 | Immediately before (10 seconds) and 1 minute after sustained passive leg raising (PLR) as well as immediately before (10 seconds) and after IV albumin infusion (total duration of procedure approximately 2 hours/patient)
  Percentage of measurements / participants where CPMX2 measurement (outcome 1) & ultrasound measurement (outcomes 3-5) are considered to be compatible, as determined by the investigator

OTHER OUTCOMES:
Assessment of Device Deficiencies (DDs), Adverse Device Effects (ADEs) and Serious Adverse Device Effects (SADEs) | During the procedure which should last about 2 hours/patient
  Safety of the procedure will be evaluated by systematically documenting Device Deficiencies (DDs), Adverse Device Effects (ADEs) and Serious Adverse Device Effects (SADEs), and by monitoring the frequency and incidence of these events (description of the adverse events, number of participants).
Identification of potential risks using the CPMX2 device | During the procedure which should last about 2 hours/patient
  Safety of the device and potential risks from using it will be assessed within the questionnaire for the practitioner and by evaluation of Device Deficiencies (description).

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Berzigotti, Prof., MD, Study Director — Insel Gruppe AG
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No